CLINICAL TRIAL: NCT04322188
Title: An Observational Study of the Use of Siltuximab (SYLVANT) in Patients Diagnosed With COVID-19 Infection Who Have Developed Serious Respiratory Complications
Acronym: SISCO
Status: Completed | Type: Observational
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Giuseppe Gritti, Principal Investigator, A.O. Ospedale Papa Giovanni XXIII
Other Study IDs: v 2 22nd April 2020
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Severe Acute Respiratory Syndrome (ARDS) Secondary to SARS-COV-2 Infection
Keywords: SARS-COV-2; ARDS; COVID-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: Patients in Cohort A were treated with siltuximab after the use of continuous positive airways pressure (CPAP) or non-invasive ventilation (NIV). Patients in Cohort B were treated after intubation
- Group 2: The control cohort will include all the patients with pneumonia/ARDS in need of non-invasive ventilation (CPAP or NIV) or intubation and not receiving experimental treatments in the ReCOVID-19-2020

INTERVENTIONS:
Other:  — this is an observational study. No intervention is applicable; patients are managed as per clinicians' best judgement and best practice

SUMMARY:
This observational study will collect data from patients treated with siltuximab program for treatment of SARS-CoV-2 infection complicated with serious respiratory complications.

This observational study will group the patients into two cohorts receiving siltuximab..

Outcome of patients will be compared to a cohort of patients receiving standard treatment without siltuximab.

The patients will be divided into 2 cohorts. Those contained in Cohort A were treated after the use of continuous positive airways pressure (CPAP) or non-invasive ventilation (NIV). Patients in Cohort B were treated after intubation

DETAILED DESCRIPTION:
This is a single-center observational cohort study that follows the use of treatment with siltuximab in patients with COVID-19 who have developed serious respiratory complications, defined by the need of ventilation (either invasive or non-invasive). Retrospective data collection will be carried out on those patients who have received siltuximab as a treatment for their Covid-19 and patients enrolled in ReCOVID19-2020, a retrospective study enrolling consecutive patients with a confirmed diagnosis of COVID-19 (interstitial pneumonia and positive test for SARS-COV-2) and who received standard treatment and who were hospitalized from 23 February up to 13 March 2020 at Papa Giovanni XXIII hospital.

The control cohort of the cohort study will include all the patients with pneumonia/ARDS in need of non-invasive ventilation (CPAP or NIV) or intubation and not receiving experimental treatments in the ReCOVID-19-2020.Patients that will be included will be divided into 2 cohorts, and per current estimation split in a 3:1 ratio: 75% will be in Cohort A as treated with CPAP/NIV, while 25% will form Cohort B and consists of patients in an ICU setting who are receiving mechanical ventilation.

Procedures outlined in this protocol are based on how the patients were managed as per clinicians' best judgement and best practice. No clinical procedures are required by this observational protocol. Data on the procedures already performed during the routine diagnosis and treatment of COVID-19 patients will be collected. The list of clinical and laboratory parameters is provided to direct data collection for this observational study (as available in the medical records).

During their hospitalization, patients will be monitored as per standard hospital practice or as per national (emergency) guidelines in accordance with extraordinary circumstances relating to the COVID-19 outbreak. After discharge, patients will be asked to provide (from their primary health care providers) relevant laboratory results and safety information for approximately 30 days following the start of COVID-19 treatment via ventilation (either mechanical or non-invasive).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and radiological diagnosis of pulmonary infection by COVID-19
2. Positive microbiological evidence of SARS-CoV-2 infection
3. Diagnosis of acute respiratory distress syndrome clinical panel in accordance with Berlin 2012 criteria
4. Need of non-invasive ventilation (NIV or CPAP) or invasive ventilation (intubation)

Exclusion Criteria:

1. Active infection of bacterial or viral (non-Covid-19) origin
2. Treatment with other anti-interleukin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The control cohort of the cohort study will include all the patients with pneumonia/ARDS in need of non-invasive ventilation (CPAP or NIV) or intubation and not receiving experimental treatments in the ReCOVID-19-2020.Patients that will be included into this observational study will be divided into 2 cohorts, and per current estimation split in a 3:1 ratio: 75% will be in Cohort A as treated with CPAP/NIV, while 25% will form Cohort B and consists of patients in an ICU setting who are receiving mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
mortality in siltuximab treated patients | 30 days
  The main objective of this study is to evaluate mortality in siltuximab treated patients and compare the results with the control cohort

SECONDARY OUTCOMES:
the need of invasive ventilation in siltuximab patients Reduction of the need of time of ventilatory support | 30 days
  Assess the need of invasive ventilation in siltuximab patients treated in cohort A and compare the results with the control cohort
clinical course of patients treated with siltuximab Percentage of patients that undergo to tracheostomy | 30 days
  Describe the clinical course of patients treated with siltuximab (Cohort A and B) in terms of ventilatory support and compare the results with the control cohort
Safety Improvement of the lung function assessed by radiologic findings | 30 days
  Safety of siltuximab treatment
the effect on inflammatory parameters | 30 days
  Evaluate the effect of siltuximab on inflammatory parameters (CRP)
Correlation of outcomes with IL-6 levels | 30 days
  Correlation of outcomes with IL-6 levels

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe GRITTI, MD, Principal Investigator — ASST PAPA GIOVANNI XXIII
Locations (1):
- ASST - Papa Giovanni XXIII, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zumla A, Hui DS, Azhar EI, Memish ZA, Maeurer M. Reducing mortality from 2019-nCoV: host-directed therapies should be an option. Lancet. 2020 Feb 22;395(10224):e35-e36. doi: 10.1016/S0140-6736(20)30305-6. Epub 2020 Feb 5. No abstract available. PMID 32035018
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452